CLINICAL TRIAL: NCT00238069
Title: Effect of CPAP (Continuous Positive Airway Pressure) on Airway Inflammation in Asthmatics With Sleep-Disordered Breathing: A Pilot Study
Brief Title: Effect of CPAP (Continuous Positive Airway Pressure) on Lung Function in Asthmatics With Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-1866
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Asthma; Sleep Apnea
Keywords: Asthma; Sleep Apnea; Obesity; CPAP
MeSH Terms: conditions — Asthma; Sleep Apnea Syndromes; Obesity

INTERVENTIONS:
Device: CPAP machine as a result of sleep study

SUMMARY:
This is a research study of asthma and sleep apnea. Our hypothesis is that untreated sleep apnea causes inflammation in the lung, which can worsen asthma. We believe treatment of sleep apnea will reduce this inflammation, and improve asthma control. This study will help us better understand what happens to the lung and bronchial tubes before and after treatment of sleep apnea, which could benefit all patients with sleep apnea. This study involves 2 bronchoscopies.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18yrs at the time of recruitment)
* Body mass index (BMI) ≥ 30
* Symptoms suggestive of sleep apnea
* Epworth Sleepiness Score (ESS) within range
* Positive sleep study for sleep apnea

Exclusion Criteria:

* Tobacco use within the last 3 months.
* Presence of other significant comorbid heart or lung disease
* Presence of another chronic inflammatory disease, such as connective-tissue disease, inflammatory bowel disease, or active infection.
* Use of systemic steroids, as defined as any prednisone use in the preceding 3 months.
* Use of leukotriene antagonists or theophylline within the preceding 6 weeks.
* Presence of severe or uncontrolled sinusitis, such that CPAP therapy will be difficult or uncomfortable.
* History of significant claustrophobia, uncontrolled psychiatric disease, or anticipated intolerance of CPAP therapy.
* Night shift workers, or other subjects with significantly altered sleep-wake cycles.
* Baseline post-bronchodilator FEV1 < 70% predicted.
* Severe gastroesophageal reflux disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-12; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Systemic inflammatory markers will include IL-6, IL-8, CRP, and TNF-α.
Exhaled breath condensate levels of IL-6 and 8-isporostane will be measured.
BAL (bronchial lavage) fluid cell count and differential, IL-6, IL-8, and TNF- α will be measured.
Endobronchial biopsies to analyze extent and type of inflammatory cell.

SECONDARY OUTCOMES:
Symptoms, albuterol use and daily morning and evening peak expiratory flows from diary cards.
Spirometry measured at three time points: before, during, and after CPAP therapy.
Post-CPAP methacholine for bronchial hyperreactivity

CONTACTS AND LOCATIONS:
Overall Officials: Richard Martin, MD, Principal Investigator — National Jewish Medical and Research Center faculty
Locations (1):
- National Jewish Medical and Research Center, Denver, Colorado, United States